CLINICAL TRIAL: NCT03349879
Title: Familial Clustering of Vitamin D Deficiency Via Shared Environment: The Korean National Health And Nutrition Examination Survey 2008-2012
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-01EXP-01-2C
Record Dates: First submitted 2017-11-16; First posted 2017-11-22 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vitamin D deficiency: serum 25(OH)D < 30 nmol/L
- Vitamin D insufficiency: serum 25(OH)D between 30 and 49 nmol/L
- Vitamin D sufficiency: serum 25(OH)D ≥ 50 nmol/L

SUMMARY:
Vitamin D deficiency is a modifiable risk factor for poor bone health. Familial correlation of serum 25-hydroxyvitamin D concentration (25(OH)D) was reported in twin- or family-based studies, mostly from Caucasian parent-offspring pairs. However, data on the familial association of 25(OH)D in extended family structure and the relative contribution of genetic and shared environmental factors on serum 25(OH)D level are limited in Asian populations. In this study, the investigators aimed to assess the relative contribution of additive genetic and environmental components on serum 25(OH)D level by variance components method in a nationwide family-based cohort. Further, the investigators will evaluate the association of vitamin D status of index individual with prevalent vitamin D deficiency of each family member including spouse, offspring, sibling, and grand-offspring. Additive influences of paternal and maternal vitamin D status on offspring will be also investigated.

DETAILED DESCRIPTION:
From the Korean National Health and Nutritional Examination Survey (KNHANES) conducted between 2008 and 2012, familial correlations for 25(OH)D will be estimated in different types of family relation pairs in 28551 subjects from 10882 families. The relative contribution of additive genetic and shared or individual environmental factors for variance of 25(OH)D level will be calculated using variance component method. Interactions between paternal and maternal vitamin D status for 25(OH)D level of offspring will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* KNHANES(Korean National Health and Nutrition Examination Survey) 2008-2012 participants

Exclusion Criteria:

* missing value on 25-hydroxyvitamin D levels
* data on another household member was unavailable
* the precise family relationship between the subjects was unclear

Ages: 10 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study was based on data from the Korean National Health and Nutrition Examination Survey (KNHANES) (IV-2, 3 and V), conducted from 2008 to 2012. The KNHANES is a nationwide cross-sectional survey performed by the Division of Chronic Disease Surveillance, Korea Centers for Disease Control and Prevention (CDC), which assessed the health, nutritional status, and socioeconomic status of the non-institutionalized civilian population of South Korea. Subjects were selected using a stratified multistage clustered probability sampling design. Families, including at least two family members with serum 25(OH)D measurements and whose family relationships could be accurately identified were selected for the study. After the selection process, a total of 28,551 subjects from 10,882 families were included in our study.
Sampling Method: Probability Sample
Enrollment: 28551 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Vitamin D deficiency | 1 minute after the survey (cross-sectional analysis)
  Vitamin D deficiency (serum 25(OH)D < 30 nmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, Department of internal Medicine, Yonsei University College of Medicine, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No